CLINICAL TRIAL: NCT02908412
Title: Evaluating and Comparing the Accuracy of Non-invasive Hemoglobin Monitoring by Spectrophotometry With and Without Digital Nerve Block in Patients Undergoing Spinal Surgery in Sina Hospital During 2016-2017
Brief Title: Non-invasive Perioperative Hb Monitoring in Spinal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: Sina Trauma and Surgery Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: IR.TUMS.VCR.REC.1395.110
Record Dates: First submitted 2016-09-15; First posted 2016-09-21 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2017-12

CONDITIONS: Blood Loss, Surgical
Keywords: Nerve Block; Spectrophotometry; Bupivacaine; Spinal Surgery; Blood Loss, Surgical
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Digital nerve block in left hand (Experimental): Patients in this group will receive DNB in left hand. DNB will be performed by injecting 2 ml of 0.25% bupivacaine at the base of medial and lateral sides of the finger attached to the sensor (1 ml on each side of the base).
  Interventions: Drug: Digital nerve block with bupivacaine
- Digital nerve block in right hand (Experimental): Patients in this group will receive DNB in right hand. DNB will be performed by injecting 2 ml of 0.25% bupivacaine at the base of medial and lateral sides of the finger attached to the sensor (1 ml on each side of the base).
  Interventions: Drug: Digital nerve block with bupivacaine

INTERVENTIONS:
Drug: Digital nerve block with bupivacaine — The aim of the study, the way it will be conducted, and the complications and possible risks are explained to them. written informed consent is obtained from them. Then, after induction of anaesthesia, an arterial line will be inserted in order to monitor blood pressure and to take blood samples. During the surgery, two rainbow adult ReSposable sensors will be attached to the third or fourth fingers of both hands, and each of sensors will be attached to a monitor. Patients will be randomly assigned to two groups: group A will receive DNB in left hand and group B will receive DNB in right hand. DNB will be performed by injecting 2 ml of 0.25% bupivacaine at the base of medial and lateral sides of the finger attached to the sensor (1 ml on each side of the base).

SUMMARY:
The decision to transfuse or not to transfuse blood products is one of the main issues in patients undergoing surgery.

The standard laboratory method of hemoglobin assessment is time-consuming, gives intermittent data, and requires venipuncture which is invasive and painful. In the past decade, the use of non-invasive and faster methods, which allow physicians to measure hemoglobin levels at the patient's bedside, have become widespread. One of the tools that make this possible is Spectrophotometric Hemoglobin.

However, one of the main concerns regarding this method is its accuracy. Since the accuracy of this assessment depends on the extent of perfusion of the organ on which the probe is placed, use of digital nerve blocks proposed to increase its accuracy.

This study aims to evaluate the effects of digital nerve block (with bupivacaine) on the accuracy of non-invasive hemoglobin monitoring by spectrophotometry in patients undergoing spinal surgery.

DETAILED DESCRIPTION:
The decision to transfuse or not to transfuse blood products is one of the main issues in healthcare systems. Timely transfusion of blood to a patient bleeding, either due to the surgery or because of the trauma, can prevent tissue hypoxia and ischemia in vital organs. However, transfusion of blood products should be done carefully and cautiously due to the potential complications of transfusions, and also because of the cost of providing blood products 1, 2, 3. Hence, during surgeries, hemoglobin level has a vital role in the diagnosis and management of patients with anemia.

The standard laboratory method of hemoglobin assessment is time-consuming, gives intermittent data, and requires venipuncture which is invasive and painful. In the past decade, the use of non-invasive and faster methods, which allow physicians to measure hemoglobin levels at the patient's bedside, have become widespread. One of the tools that make this possible is Spectrophotometric Hemoglobin (SpHb Masimo Rainbow Co-oximeter). This procedure is applied by a digital probe and allows physicians to monitor hemoglobin levels continuously. 4, 5, 6 However, one of the main concerns regarding this method is its accuracy. Actually, the difference between the measured hemoglobin level and the actual hemoglobin level of the patient, might make it impossible for physicians to decide with sufficient confidence3.

From the time that SpHb has been available in operating rooms, various studies have evaluated its accuracy. While its accuracy has been reported relatively acceptable (mean difference is about 1-1.5 g/dl comparing to the lab data),4 there are still concerns regarding this issue. Furthermore, it is not clear whether this difference would remain the same during the surgery or not. Because blood transfusion is rarely needed when the hemoglobin level of patient is higher than 10g/dl during the surgery. Also, blood transfusion becomes obviously necessary if hemoglobin levels drop to 6g/dl or lower during the surgery. Therefore, the accuracy of the tool in assessing hemoglobin levels at this critical interval (6-10g/dl) is of greater importance.6,7 Experimental studies have confirmed that accuracy could change in different hemoglobin levels5,8, and with the passage of time.9 In addition, it has been reported that after significant blood loss or even following injection of blood, the average difference between SpHb and laboratory might change, as well. 5,8 Since the accuracy of this assessment depends on the extent of perfusion of the organ on which the probe is placed, methods that enhance blood circulation in the organ (including local heating of the organ and use of digital nerve blocks (DNB), proposed to increase its accuracy.10, 11 In a study conducted in 2012 by Miller et al. on 20 patients undergoing spinal surgery, DNB was performed using lidocaine. The differences between SpHb and lab hemoglobin were recorded first after injection, and then at almost hourly intervals. These differences were compared to data from another study without DNB. Thirty seven percent of data in the intervention group and 12% of data in the control group was considered as "very accurate". Results of this study showed that DNB increased perfusion indices and SpHb accuracy.10 Following the previous study, Miller et al. carried out a study in 2014 to compare the effects of DNB with lidocaine and bupivacaine on 12 healthy volunteers. DNB was performed on two identical fingers on both hands of the volunteers. Lidocaine was used on one hand and bupivacaine on the other one. Results of this study showed that both lidocaine and bupivacaine raised the perfusion indices and temperatures of the fingers. The duration and extent of the rise in temperature were more for bupivacaine, and there was a direct correlation between changes in perfusion index and those in SpHb.11 Since, the previous study data had been gathered from healthy individuals, this study aims at investigate the effects of DNB on the accuracy SpHb in patients undergoing surgery.

ELIGIBILITY:
Inclusion Criteria: All patients 18 years of age or older, admitted to Sina hospital to have spinal surgery, whose surgery is not an emergency, are included in the study. Moreover, the patients must be in grade 2 or lower according to the ASA Physical Status Classification, and volunteer to participate in the study.

-

Exclusion Criteria: Patients who are going to have an emergency surgery are excluded from the study. Also patients with grade 3 ASA or higher, or the ones suffering from anatomic or vascular disorders that cause problems in attaching the SpHb sensor, are excluded from the study.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
accuracy of SpHb | At the start of the operation, once every 1.5 hours during the operation till its end
  in each patient, Sphb values will be documented for both hands. Also, the arterial blood sample (lab Hb) will be sent to the laboratory. The difference between two measure in each hand (with or without DNB) shows the accuracy of Sphb for each hand.

SECONDARY OUTCOMES:
Perfusion index (PI) | At the start of the operation, once every 1.5 hours during the operation till its end
  In each patient, PI value of hand with DNB will be compared to PI measure in the other hand.
Pleth Variability Index (PVI) | At the start of the operation, once every 1.5 hours during the operation till its end
  In each patient, PVI value of hand with DNB will be compared to PI measure in the other hand.

CONTACTS AND LOCATIONS:
Locations (1):
- Sina Hospital, Tehran, Tehtan, Iran

REFERENCES:
- [Background] Barker SJ, Shander A, Ramsay MA. Continuous Noninvasive Hemoglobin Monitoring: A Measured Response to a Critical Review. Anesth Analg. 2016 Feb;122(2):565-72. doi: 10.1213/ANE.0000000000000605. PMID 25746056
- [Background] Lamhaut L, Apriotesei R, Combes X, Lejay M, Carli P, Vivien B. Comparison of the accuracy of noninvasive hemoglobin monitoring by spectrophotometry (SpHb) and HemoCue(R) with automated laboratory hemoglobin measurement. Anesthesiology. 2011 Sep;115(3):548-54. doi: 10.1097/ALN.0b013e3182270c22. PMID 21716091
- [Background] Suehiro K, Joosten A, Alexander B, Cannesson M. Continuous noninvasive hemoglobin monitoring: ready for prime time? Curr Opin Crit Care. 2015 Jun;21(3):265-70. doi: 10.1097/MCC.0000000000000197. PMID 25827587
- [Background] Kim SH, Lilot M, Murphy LS, Sidhu KS, Yu Z, Rinehart J, Cannesson M. Accuracy of continuous noninvasive hemoglobin monitoring: a systematic review and meta-analysis. Anesth Analg. 2014 Aug;119(2):332-346. doi: 10.1213/ANE.0000000000000272. PMID 24914627
- [Background] Applegate RL 2nd, Barr SJ, Collier CE, Rook JL, Mangus DB, Allard MW. Evaluation of pulse cooximetry in patients undergoing abdominal or pelvic surgery. Anesthesiology. 2012 Jan;116(1):65-72. doi: 10.1097/ALN.0b013e31823d774f. PMID 22133758
- [Background] Rice MJ, Gravenstein N, Morey TE. Noninvasive hemoglobin monitoring: how accurate is enough? Anesth Analg. 2013 Oct;117(4):902-907. doi: 10.1213/ANE.0b013e31829483fb. Epub 2013 Jul 10. PMID 23842195
- [Background] Giraud B, Frasca D, Debaene B, Mimoz O. Comparison of haemoglobin measurement methods in the operating theatre. Br J Anaesth. 2013 Dec;111(6):946-54. doi: 10.1093/bja/aet252. Epub 2013 Jul 17. PMID 23869108
- [Background] Park YH, Lee JH, Song HG, Byon HJ, Kim HS, Kim JT. The accuracy of noninvasive hemoglobin monitoring using the radical-7 pulse CO-Oximeter in children undergoing neurosurgery. Anesth Analg. 2012 Dec;115(6):1302-7. doi: 10.1213/ANE.0b013e31826b7e38. Epub 2012 Nov 9. PMID 23144437
- [Background] Miller RD, Ward TA, Shiboski SC, Cohen NH. A comparison of three methods of hemoglobin monitoring in patients undergoing spine surgery. Anesth Analg. 2011 Apr;112(4):858-63. doi: 10.1213/ANE.0b013e31820eecd1. Epub 2011 Mar 8. PMID 21385985
- [Background] Miller RD, Ward TA, McCulloch CE, Cohen NH. Does a digital regional nerve block improve the accuracy of noninvasive hemoglobin monitoring? J Anesth. 2012 Dec;26(6):845-50. doi: 10.1007/s00540-012-1452-0. Epub 2012 Aug 1. PMID 22850903
- [Background] Miller RD, Ward TA, McCulloch CE, Cohen NH. A comparison of lidocaine and bupivacaine digital nerve blocks on noninvasive continuous hemoglobin monitoring in a randomized trial in volunteers. Anesth Analg. 2014 Apr;118(4):766-71. doi: 10.1213/ANE.0000000000000144. PMID 24651230